CLINICAL TRIAL: NCT01591967
Title: A Randomized Controlled Trial to Measure the Effects of Specific Thoracic Chiropractic Adjustments on Blood Pressure and Pulse Rate
Brief Title: Measure the Effects of Specific Thoracic Chiropractic Adjustments on Blood Pressure and Pulse Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spinal Missions, Inc., LLC (Other)
Responsible Party: Principal Investigator, Dr. Steven D. Roffers, Director of Research, Spinal Missions, Inc., LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM001
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension
Keywords: Chiropractic; Blood pressure; Pulse Rate; Thoracic
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Control -- no intervention
- Placebo w/ sham (No Intervention): Sham intervention with the adjusting tool turned "off"
- Activator treatment (Experimental): Treatment with Activator
  Interventions: Device: Activator IV Adjusting Instrument

INTERVENTIONS:
Device: Activator IV Adjusting Instrument — Activator (http://www.activator.com/products-page/) adjustment effects on BP and PR
  Other Names: Activator adjusting instrument; http://www.activator.com/products-page/
  Arms: Activator treatment

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to measure the effects of specific thoracic (T5 to T1) chiropractic adjustments on BP and PR in a larger sample size of both normotensive and hypertensive humans.

DETAILED DESCRIPTION:
OBJECTIVE: Previous studies on the effects of chiropractic treatment on blood pressure (BP) and pulse rate (PR) have reported decreases in both systolic and diastolic BP, as well as PR. However, many of those studies have been criticized for various study flaws, and accused of drawing erroneous conclusions, due to small sample size and various methodological concerns. The purpose of this randomized controlled trial (RCT) is to measure the effects of specific thoracic (T5 to T1) chiropractic adjustments on BP and PR in a larger sample size of both normotensive and hypertensive humans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were invited to participate in accordance with the Guidelines for Chiropractic Quality Assurance and Practice Parameters: proceedings of the Mercy Center Consensus Conference, Gaithersburg, MD, 1993, Aspen Publishers Inc.

Additionally and specifically for this RCT:

1. Both male and female subjects age 18 years and older were invited to participate
2. Subjects must not be pregnant
3. Subjects must not have any recent or current fractures of the arms or legs
4. Subjects must not have any visceral or abdominal condition such that being in the prone position would be detrimental to their health
5. Subjects must not have any known primary cancers of the spine or spinal column, nor any secondary metastatic process of the spine or spinal column
6. Subjects must not be under the influence of drugs or alcohol
7. Subjects must not have vertigo or any other imbalance condition
8. Subjects must not have any arm or leg prosthetic device
9. Subjects must be able to understand spoken and/or written Spanish and/or English

Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The purpose of this randomized controlled trial (RCT) was to measure the effects of specific thoracic (T5 to T1) chiropractic adjustments on BP and PR in a larger sample size of both normotensive and hypertensive humans. | Baseline, pre-adjustment, post-adjustment
  OBJECTIVE: Previous studies on the effects of chiropractic treatment on blood pressure (BP) and pulse rate (PR) have reported decreases in both systolic and diastolic BP, as well as PR. However, many of those studies have been criticized for various study flaws, and accused of drawing erroneous conclusions, due to small sample size and various methodological concerns. The purpose of this randomized controlled trial (RCT) was to measure the effects of specific thoracic (T5 to T1) chiropractic adjustments on BP and PR in a larger sample size of both normotensive and hypertensive humans.

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Roffers, DC, Principal Investigator — Spinal Missions, Inc., LLC